CLINICAL TRIAL: NCT05421689
Title: A Multi-Center, Double-Blind, Randomized Placebo-Controlled Investigation of Autologous Muscle Derived Cells (AMDC) for the Treatment of Tongue Dysphagia Resulting From the Treatment of Head and Neck Cancer
Brief Title: Autologous Muscle Derived Cells for Treatment of Tongue Dysphagia
Acronym: REVIVE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1800521; 1800521 (Other: UC DAVIS)
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, multicenter clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will receive two treatments of intramuscular injection of 1 AMDC-GIR dose of 150 x 10⁶ cells or identical placebo. Both patients and study investigators at all sites will be blinded to the treatment assignment of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: 150 x 10⁶ AMDC-GIR dosage (Experimental): 33 subjects will be receiving two doses of 150 x 10⁶ AMDC-GIR spaced 4-6 weeks apart.
  Interventions: Biological: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR)
- Experimental: Identical Placebo composed of the same cryopreservation medium used for AMDC-GIR (Sham Comparator): 33 subjects will be receiving two doses of identical placebo composed of the same cryopreservation medium used for AMDC-GIR. Doses will be spaced 4-6 weeks apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) — The study will treat 66 patients at 2 clinical sites: UC Davis Center for Voice and Swallowing and UCSF Voice and Swallowing Center. Patients will be randomized 1:1 to receive either 2 AMDC-GIR doses of 150 x 10⁶ cells or 2 doses of identical placebo composed of the same cryopreservation medium used for AMDC-GIR. Enrollment is expected to be completed within 2 years of initiating the study. Patients will be followed for 24 months post-treatment.
  Other Names: Autologous muscle derived stem cells
  Arms: Experimental: 150 x 10⁶ AMDC-GIR dosage
Other: Placebo — two doses of placebo will be administered and spaced 4-6 weeks apart.
  Other Names: identical placebo composed of the same cryopreservation medium used for AMDC-GIR
  Arms: Experimental: Identical Placebo composed of the same cryopreservation medium used for AMDC-GIR

SUMMARY:
The primary objective of this double-blind, randomized, placebo-controlled, multicenter clinical trial is to evaluate the safety of AMDC-GIR during the 24 months following 2 consecutive treatments of tongue dysphagia in male and female patients who have undergone surgery and/or chemo- and/or radiotherapy for squamous cell cancer of the oropharynx.

DETAILED DESCRIPTION:
The purpose of this double-blind, randomized, placebo-controlled, multicenter clinical trial is to evaluate the safety and efficacy of Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) for the treatment of tongue dysphagia (TD) in male and female patients who have undergone surgery and/or chemo- and/or radiotherapy for squamous cell cancer of the oropharynx.

Surgery, chemo- and radiotherapy induce significant TD and result in long-term swallowing dysfunction. The incidence of TD after treatment for cancer of the pharynx exceeds 80%. Therefore, augmenting tongue muscle function may be beneficial to patients. Autologous muscle cell therapy, which involves isolation of cells from skeletal muscle biopsies, ex vivo expansion, and subsequent injection into the tongue, may serve as a durable therapy. In animal studies, muscle derived cells have successfully integrated within tissue to improve tongue strength and function. Intramuscular injection of AMDC-GIR has been shown to produce localized tissue changes at the injection site without a systemic effect. Initial results of a Phase 1 open label trial suggest that 150 x 10⁶ AMDC-GIR for the treatment of TD is safe and may be efficacious. A Phase I/II placebo controlled, randomized clinical trial is warranted.

Patients will receive two treatments of intramuscular injection of 1 AMDC-GIR dose of 150 x 10⁶ cells or identical placebo. For entrance into the study, patients must meet the study inclusion criterion and must not meet any of the exclusion criteria. Patients will have quantitative and qualitative measures of swallowing impairment assessed before treatment and at prescheduled intervals after treatment.

The study will treat 66 patients at 2 clinical sites: UC Davis Center for Voice and Swallowing and UCSF Voice and Swallowing Center. Patients will be randomized 1:1 to receive either 2 AMDC-GIR doses of 150 x 10⁶ cells or 2 doses of identical placebo composed of the same cryopreservation medium used for AMDC-GIR. Enrollment is expected to be completed within 2 years of initiating the study. Patients will be followed for 24 months post-treatment.

Male and female patients at least 18 years of age who have undergone surgery and/or chemo- and/or radiotherapy for primary treatment of oropharyngeal squamous cell cancer and who present with symptoms and findings of TD will be eligible for participation. Eligible patients will have muscle tissue harvested using an established needle biopsy technique during an outpatient procedure.

The harvested muscle will be placed in a hypothermic medium and transported to the manufacturer for cell processing. The muscle derived cells (MDC) will be isolated and expanded in culture over several weeks to a final AMDC-GIR dose of 150 x 10⁶ cells. Each patient will receive 2 doses of cells or placebo spaced 4-6 weeks apart.

After reaching the desired concentration, the isolated and expanded AMDC-GIR or identical placebo will be frozen and shipped back to the investigating physician. The investigative team will thaw the AMDC-GIR and dilute the sample with an equal volume of physiological saline. Under direct vision, the resulting suspension will be injected into the patient's tongue in a brief outpatient procedure for the patients randomized to the treatment arm. Patients randomized to receive placebo will undergo an identical procedure utilizing a thawed solution of frozen media without cells. Both patient and clinician will be blind to the treatment and placebo status.

Patients will be assessed for improvement in TD at 6 months, 12 months and 18 months and 24 months following treatment. Adverse events will be assessed at those visits, as well as during virtual visits at 1-2 days, 1 week, 4 weeks, 3 months, 15 months, 21 months and 24 months. Adverse events will also be assessed at 6 months post-injection in patients who were in the placebo group and elected to receive AMDC_GIR injections after the unblinding. Patient reported outcome measures will be assessed at 4 weeks, 3 months, 6 months, 12 months, 18 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, at least 18 years old, with primary symptoms of TD following surgery and/or chemo- and/or radiotherapy for treatment of squamous cell carcinoma for oropharyngeal cancer. Treatment must be completed at least 24 months prior to enrollment, with TD and disease-free status confirmed by medical history, clinical symptoms, a focused head and neck examination, swallowing fluoroscopy, and high-resolution pharyngeal manometry.
2. TD severity should be moderate as defined by a Functional Oral Intake Scale (FOIS, provided in Appendix C). Individuals must have a FOIS of 3 or better and EAT-10 score of greater than 5.
3. Patient has failed to achieve resolution of symptoms following contemporary therapies.

Exclusion Criteria:

1. Simultaneously participating in another investigational drug or device study or has completed the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
2. Previously treated with an investigational device, drug, or procedure for TD within 6 months prior to signing consent.
3. TD of neurogenic etiology or uncorrected congenital abnormality leading to TD.
4. Neuromuscular disorder (e.g., Parkinson's disease, muscular dystrophy, multiple sclerosis) that could lead to TD.
5. Severe fibrosis at injection site.
6. Uncontrolled diabetes.
7. Compromised immune system due to disease state, chronic corticosteroid use, or other immunosuppressive therapy.
8. Medical condition or disorder that may limit life expectancy or that may cause CIP deviations (e.g., unable to perform self-evaluations or accurately report medical history, symptoms, or data).
9. History of bleeding diathesis or uncorrectable coagulopathy.
10. Known allergy or hypersensitivity to bovine proteins or allergens, gentamicin sulfate, or ampicillin that medically warrants exclusion as determined by the physician.
11. Any non-skin cancer that has necessitated treatment within the past 24 months.

Patient's Current Status-based Criteria:

1. Evidence or known high risk of recurrent or persistent cancer as determined by the physician during screening.
2. Tests positive for Hepatitis B (required tests: Hepatitis B Surface Antigen [HBsAg] and Anti-Hepatitis B Core Antibody [Anti-HBc]), Hepatitis C (required test: Hepatitis C Antibody [Anti-HCV]), HIV (required tests: HIV Type 1 and 2 Antibodies [Anti-HIV-1, 2]), and/or Syphilis.

   a. Tests performed by certified/authorized testing laboratory using licensed/approved tests and performed on blood samples collected within 30 days prior to muscle tissue procurement.
3. Cannot, or is not willing to maintain the current treatment regimen for existing contemporary therapy (e.g., swallowing therapy).
4. Requires prophylactic antibiotics for chronic infection or has required 2 or more courses of antibiotics for infections in the 2 months prior to signing consent.
5. Any condition, including current infection or immunodeficiency, which could lead to significant postoperative complications.
6. Refuses or cannot provide written informed consent.
7. Not available for, or willing to comply with the baseline and follow-up evaluations as required by the CIP.
8. Pregnant, lactating, or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Study product-related, biopsy procedure-related, and injection procedure-related adverse events. | 24 months
  Safety will be determined by the frequency and severity of adverse events related to study procedures and study product.
Anterior tongue pressure measured from Iowa Oral Performance Instrument (IOPI) | 24 months
  Efficacy of AMDC-GIR in the improvement of objective Anterior Tongue Pressure Measurement (IOPI)

SECONDARY OUTCOMES:
Incidence of patient aspiration pneumonia | 24 months
  Effects of AMDC-GIR on incidence of patient reported aspiration pneumonia (yes/no scoring criteria)
Incidence of patient survival | 24 months
  Effects of AMDC-GIR on incidence of patient reported survival (yes/no scoring criteria)
Penetration Aspiration scale rating following swallowing fluoroscopy | 24 months
  The 8-point Penetration-Aspiration Scale (scores of 1-8, 1=better, 8=worse, see table below) is the standard method used measure the severity of airway invasion during swallowing.
  1. Material does not enter the airway
  2. Material enters the airway, remains above the vocal folds, and is ejected from the airway
  3. Material enters the airway, remains above the vocal folds, and is not ejected from the airway
  4. Material enters the airway, contacts the vocal folds, and is ejected from the airway
  5. Material enters the airway, contacts the vocal folds, and is not ejected from the airway
  6. Material enters the airway, passes below the vocal folds, and is ejected into the larynx or out of the airway
  7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort
  8. Material enters the airway, passes below the vocal folds, and no effort is made to eject
Peak Pharyngeal pressure measurement from high-resolution manometry | 24 months
  Efficacy of AMDC-GIR in the improvement of objective manometric swallowing parameters
Patient-reported dysphagia symptoms based on Eating Assessment Tool EAT10 score | 24 months
  Survey consisting of 10 questions (see table below), each score on a scale of 0-4, with 0= no problem, 4= severe problem.
  922 Belafsky et al. Eating Assessment Tool TABLE 3. EATING ASSESSMENT TOOL (EAT-10) Circle the appropriate response. To what extent are the following scenarios problematic for you?
  1. My swallowing problem has caused me to lose weight.
  2. My swallowing problem interferes with my ability to go out for meals.
  3. Swallowing liquids takes extra effort.
  4. Swallowing solids takes extra effort.
  5. Swallowing pills takes extra effort.
  6. Swallowing is painful.
  7. The pleasure of eating is affected by my swallowing.
  8. When I swallow food sticks in my throat.
  9. I cough when I eat.
  10. Swallowing is stressful

OTHER OUTCOMES:
Pharyngeal Constriction Ratio measurement for swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Upper Esophageal Sphincter opening measurement for swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Pharyngeal transit time measurement for swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Patient-reported survey of smell and taste | 24 months
  Effects of AMDC-GIR on patient reported smell and taste as reported by the 8-question survey ChemoSensory Questionnaire (CCQ). Minimum score for each scale, 4 Maximum score for each scale, 20. High score indicates better function
Clinical assessment of vocal quality (CAPE-V) | 24 months
  Effects of AMDC-GIR in the improvement of objective voice quality. The CAPE-V approach uses a form where Overall Severity, Roughness, Breathiness, Strain, Pitch, and Loudness are rated using a 100-mm visual analog scale. The rater places a vertical mark along each horizontal line where the far left end of the line represents the least impaired status and the far right represents the one most impaired. Scores are obtained by making measurements to the nearest millimeter from the left most (least impaired) end of the horizontal line. The higher the score the worse the impairment.
Patient-reported Quality of Life based on FACT-HN score | 24 months
  Effects of AMDC-GIR on patient reported quality of life. FACT-HN is a 39-question survey, with a score range from 0-148. The higher the score the better the quality of life for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, Principal Investigator — University of California Davis, Department of Otolaryngology; Maggie Kuhn, MD, Principal Investigator — University of California Davis, Department of Otolaryngology; Johnathon D Anderson, PhD, Study Director — University of California Davis, Department of Otolaryngology
Locations (2):
- United States (2):
  - UC Davis Medical Center, Department of Otolaryngology, Sacramento, California
  - UC San Francisco Medical Center, Voice and Swallow Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No